CLINICAL TRIAL: NCT01410942
Title: Multimodal Therapy for the Treatment of Fatigue in Patients With Prostate Cancer Receiving Radiotherapy With Androgen Deprivation Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-0389; RSG-11-170-01-PCSM (Other: Amercian Cancer Society); NCI-2011-02764 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Multimodal Therapy; MMT; Fatigue; Cognitive Behavioral Therapy; CBT; Radiation therapy; Radiotherapy; RT; Functional Assessment of Chronic Illness Therapy - Fatigue; FACIT-F; Androgen deprivation therapy; Methylphenidate; Methylphenidate Hydrochloride; Ritalin; Concerta; Placebo; Sugar Pill
MeSH Terms: conditions — Prostatic Neoplasms; Fatigue | interventions — Sugars; Methylphenidate; Counseling; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Placebo + Sham Exercise (Placebo Comparator): Placebo capsules by mouth twice daily. Participants in sham exercise intervention meet with exercise physiologist in person on first visit to learn stretching exercises and receive written instructions same as those receiving exercise therapy.
  Interventions: Other: Placebo; Behavioral: Counseling Sessions; Other: Sham Exercise
- Methylphenidate + Sham Exercise (Experimental): Methylphenidate starting dose 5 mg by mouth twice daily. Participants in sham exercise intervention meet with exercise physiologist in person on first visit to learn stretching exercises and receive written instructions same as those receiving exercise therapy.
  Interventions: Drug: Methylphenidate; Behavioral: Counseling Sessions; Other: Sham Exercise
- Exercise + Placebo (Placebo Comparator): Resistance exercise sessions completed 3 days a week allowing at least 48 hours between each session, and walk minimum of 5 days a week at intensity and duration established by exercise physiologist. Placebo capsules by mouth twice daily.
  Interventions: Other: Placebo; Behavioral: Counseling Sessions; Other: Standardized Exercise Intervention Program
- Cognitive Therapy + Placebo (Placebo Comparator): Cognitive Therapy - 8 weekly sessions (1 in person and 7 by telephone) lasting 45 minutes each, during which review learned relaxation skills and taught new cognitive and/or behavioral skill. Placebo capsules by mouth twice daily.
  Interventions: Other: Placebo; Other: Sham Exercise; Other: Cognitive Behavioral Therapy (CBT)
- Methylphenidate + Exercise (Experimental): Methylphenidate starting dose 5 mg by mouth twice daily. Resistance exercise sessions completed 3 days a week allowing at least 48 hours between each session, and walk minimum of 5 days a week at intensity and duration established by exercise physiologist.
  Interventions: Drug: Methylphenidate; Behavioral: Counseling Sessions; Other: Standardized Exercise Intervention Program
- Methylphenidate + Cognitive Therapy (Experimental): Methylphenidate starting dose 5 mg by mouth twice daily. Cognitive Therapy - 8 weekly sessions (1 in person and 7 by telephone) lasting 45 minutes each, during which review learned relaxation skills and taught new cognitive and/or behavioral skill.
  Interventions: Drug: Methylphenidate; Other: Sham Exercise; Other: Cognitive Behavioral Therapy (CBT)
- Exercise + Cognitive Therapy + Placebo (Placebo Comparator): Resistance exercise sessions completed 3 days a week allowing at least 48 hours between each session, and walk minimum of 5 days a week at intensity and duration established by exercise physiologist. Cognitive Therapy - 8 weekly sessions (1 in person and 7 by telephone) lasting 45 minutes each, during which review learned relaxation skills and taught new cognitive and/or behavioral skill. Placebo capsules by mouth twice daily
  Interventions: Other: Placebo; Other: Standardized Exercise Intervention Program; Other: Cognitive Behavioral Therapy (CBT)
- Methylphenidate + Exercise + Cognitive Therapy (Experimental): Methylphenidate starting dose 5 mg by mouth twice daily. Resistance exercise sessions completed 3 days a week allowing at least 48 hours between each session, and walk minimum of 5 days a week at intensity and duration established by exercise physiologist. Cognitive Therapy - 8 weekly sessions (1 in person and 7 by telephone) lasting 45 minutes each, during which review learned relaxation skills and taught new cognitive and/or behavioral skill.
  Interventions: Drug: Methylphenidate; Other: Standardized Exercise Intervention Program; Other: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Other: Placebo — Capsules by mouth twice daily.
  Other Names: sugar pill
  Arms: Cognitive Therapy + Placebo; Exercise + Cognitive Therapy + Placebo; Exercise + Placebo; Placebo + Sham Exercise
Drug: Methylphenidate — Starting dose 5 mg by mouth twice daily.
  Other Names: Methylphenidate Hydrochloride; Ritalin; Concerta
  Arms: Methylphenidate + Cognitive Therapy; Methylphenidate + Exercise; Methylphenidate + Exercise + Cognitive Therapy; Methylphenidate + Sham Exercise
Behavioral: Counseling Sessions — 8 weekly sessions (1 in person and 7 by telephone) lasting 45 minutes each.
  Other Names: Counseling
  Arms: Exercise + Placebo; Methylphenidate + Exercise; Methylphenidate + Sham Exercise; Placebo + Sham Exercise
Other: Sham Exercise — Participants in placebo/sham exercise intervention meet with exercise physiologist in person on first visit to learn stretching exercises and receive written instructions same as those receiving exercise therapy.
  Arms: Cognitive Therapy + Placebo; Methylphenidate + Cognitive Therapy; Methylphenidate + Sham Exercise; Placebo + Sham Exercise
Other: Standardized Exercise Intervention Program — Resistance exercise sessions completed 3 days a week allowing at least 48 hours between each session, and walk minimum of 5 days a week at intensity and duration established by exercise physiologist.
  Arms: Exercise + Cognitive Therapy + Placebo; Exercise + Placebo; Methylphenidate + Exercise; Methylphenidate + Exercise + Cognitive Therapy
Other: Cognitive Behavioral Therapy (CBT) — 8 weekly sessions (1 in person and 7 by telephone) lasting 45 minutes each, during which review learned relaxation skills and taught new cognitive and/or behavioral skill.
  Arms: Cognitive Therapy + Placebo; Exercise + Cognitive Therapy + Placebo; Methylphenidate + Cognitive Therapy; Methylphenidate + Exercise + Cognitive Therapy

SUMMARY:
The goal of this clinical research study is to learn about the effect of different combinations of exercise, supportive counseling, and methylphenidate/placebo for the treatment of fatigue in patients with prostate cancer. The safety of this treatment combination will also be studied.

Methylphenidate is a stimulant designed to increase the activity of the central nervous system.

A placebo is not a drug. It looks like the study drug but is not designed to treat any symptom, disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

The exercise in this study is designed to help improve your physical fitness and energy levels.

Supportive counseling is designed to help to control symptoms, fatigue, anxiety, depression, pain, and/or sleep disorders.

DETAILED DESCRIPTION:
If you are found eligible and agree to take part in the study:

* You will complete a baseline exercise assessment which will last about 30-45 minutes and include the following:
* A sit-to-stand test. You will sit in chair with your arms across your chest. Then you will be timed as you stand and sit down 5 times as quickly as possible.
* A hand-grip strength test. You will grip a device with each hand as hard as you can.
* A 6-minute walk test. You will be timed while you walk on a 100-foot loop. You will walk 50 feet and then turn and walk back to the beginning. You will do this at a walking speed that feels comfortable and for as many times as you can in 6 minutes.
* You will be given a belt (accelerometer) that you are required to wear for the first week of treatment. The accelerometer measures your physical activity.

Study Groups:

You will be randomly assigned (as in the roll of dice) to 1 of 8 study groups. You will have an equal chance of being assigned to any group. You will have a 50% chance of receiving the placebo.

The exercises and skills learned during counseling will be different for each study group. The study staff will talk to you about your assigned exercises and skills. You will be assigned to 1 of 2 types of exercise groups. One group will do resistance exercises and walking, and the other group will do stretching.

You be assigned to 1 of 2 types of counselling groups. One group will receive education on relaxation and symptoms. The other group will receive standard supportive counseling.

Neither you nor the medical study staff will know which group you are in. Only the study staff who will work with you for the exercise and counseling will know which group you are in. If needed for your safety, the medical staff will be able to find out which group you are in.

Study Drug/Placebo Administration:

You will take the methylphenidate/placebo capsules by mouth with water, 2 times each day. You must take both doses before 3 PM and wait at least 2 hours between doses.

Study Visits:

For all study visits/calls, you will be asked about any drugs you may be taking or any side effects that you may be having. At home during the study, you will continue practicing exercises from the exercise sessions and skills from the counseling sessions.

On Day 1, if not done at Screening:

* Your medical history will be recorded.
* You will have a physical exam, including measurement of your vital signs.
* You will complete 5 questionnaires, which should last about 30 minutes. The questionnaires ask about:
* Your emotional and physical well being
* Your level of fatigue
* Any anxiety and/or depression you may be having
* Any symptoms you may be having

On Day 8 (+/- 3 days):

* You will meet with a counselor. You will be asked to discuss your thoughts and feelings on different topics related to your well-being. The counseling session will last about 45 minutes.
* You will meet with the exercise trainer. The exercise trainer will teach you exercises and give you written instructions for how to do them at home. The exercise meeting will last about 30-45 minutes.
* You will be asked to complete a questionnaire that asks about any symptoms and/or side effects that you may be having. This should take about 10 minutes.

On Days 15 and 29 (+/- 3 days):

* You will exercise and then be asked how the exercises are going either in person or later over the phone. This should last about 30 minutes.
* You will have a counseling session with a counselor over the phone. This should last about 45 minutes.
* You will complete the 5 questionnaires.

On Days 22 and 36 (+/- 3 days) the exercise trainer and the counselor will call. These calls should last between 30-45 minutes.

On Day 43 (+/- 3 days) the exercise trainer and the counselor will call. These calls should last between 30-45 minutes.

-You will complete a questionnaire that asks about any symptoms and/or side effects you may be having. This should take about 10 minutes.

On Day 50 (+/- 3 days) the exercise trainer and the counselor will call if you have any uncompleted sessions. These calls should last between 30-45 minutes.

-You will be given an accelerometer that you are required to wear for the last week of treatment.

On Day 57 (+/- 10 days) you will return to the clinic:

* You will have a physical exam, including measurement of your vital signs.
* You will complete a sit-to-stand test.
* You will complete a hand-grip strength test.
* You will complete a 6-minute walk test.
* You will complete the 5 questionnaires.

Length of Study Participation:

You may continue taking the study drug/placebo for up to 57 days (+/- 10 days). You will no longer be able to take the study drug/placebo if the disease gets worse, if intolerable side effects occur, if you are unable to follow study directions, or if you cannot complete enough of the treatment combination as planned.

Your participation on the study will be over after you have completed the follow-up visit.

Follow-Up Visit:

About 3 months after your last dose of study drug/placebo, you will return to the clinic for a follow-up visit:

* You will be asked about any side effects you may have had.
* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* You will complete a sit-to-stand test.
* You will complete hand-grip strength tests.
* You will complete a 6-minute walk test.
* You will be asked to complete the 5 questionnaires.

This is an investigational study. Methylphenidate tablets are FDA approved and commercially available for the treatment of attention deficit disorder (ADD). The methylphenidate capsules made from the methylphenidate tablets especially for this study are not approved by the FDA. The combination of methylphenidate, exercise, and counseling is considered investigational.

Up to 175 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of prostate cancer and are scheduled to receive radiotherapy with androgen deprivation therapy
2. Rate fatigue at least 1 or higher on a scale of 0-10.
3. Describe fatigue as being present every day for most of day for a minimum of 2 weeks.
4. Have no clinical evidence of cognitive failure as evidenced by Memorial Delirium Assessment Scale (MDAS) score of </=13 at baseline.
5. Be aged 18 years or older.
6. Be willing to engage in follow-up telephone calls with a research nurse/coordinator.
7. Be willing to participate in the exercise and in Cognitive Behavioral Therapy (CBT).
8. Have telephone access to be contacted by the research nurse/coordinator.
9. Have a hemoglobin level of >/=10 g/dL within 2 weeks of enrollment.
10. Be able to understand the description of the study and give written informed consent.
11. Have a Zubrod performance status of 0 to 2.

Exclusion Criteria:

1. Have a major contraindication to MP (e.g., allergy/hypersensitivity to study medications or their constituents), exercise (e.g., cardiac disease), cognitive behavioral therapy (e.g., schizophrenia), or conditions making adherence difficult as determined by the attending physician.
2. Be currently taking MP or have taken it within the previous 10 days.
3. Are regularly engaged in moderate- or vigorous-intensity exercise for at least 150 minutes per week.
4. Regularly used cognitive behavioral therapy in the last 6 weeks.
5. Be unable to complete the baseline assessment forms or to understand the recommendations for participation in the study.
6. Need monoamine oxidase inhibitors, tricyclic antidepressants, or clonidine.
7. Have glaucoma.
8. Have with history of severe cardiac disease (New York Heart Association functional class III or IV).
9. Have tachycardia and/or uncontrolled hypertension
10. Be currently receiving anticoagulants, anticonvulsants (phenobarbital, diphenylhydantoin, primidone), phenylbutazone, and/or tricyclic drugs (imipramine, clomipramine, or desipramine).
11. History of uncontrolled hypothyroidism as evidenced by thyroid test (TSH) within the last month, hypercalcemia or hyperglycemia (within the last 15 days).
12. Unable to speak and understand English
13. Any medical or psychological condition or any reason that, according to the investigator's judgment, makes the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2012-02-08 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) subscale scores | Baseline and on Day 57
  Effects of various treatments[exercise, Cognitive Behavioral Therapy (CBT), Methylphenidate] and combinations of treatments in Multimodal Therapy (MMT) in reducing cancer-related fatigue in participants with prostate cancer receiving radiotherapy (RT), as measured by change in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) subscale scores taken at baseline and on Day 57.

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennurajalingam, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org